CLINICAL TRIAL: NCT05289570
Title: A Phase 2b Open-Label, Single Arm Study to Evaluate the Efficacy of Voxelotor for Improving Oxygen Saturation and Reducing Ventilatory Support Requirements in Adult Patients With New or Increased Oxygen Requirement
Brief Title: Voxelotor for Improving Oxygen Saturation in Adults
Acronym: Voxelotor
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated by new sponsor due to funding issues.
Sponsor: Duke University (Other)
Responsible Party: Principal Investigator, Ian Welsby, MD, Principal Investigator, Duke University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00109353
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Results first posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-06

CONDITIONS: Acute Lung Injury; End Stage Lung Disease
MeSH Terms: conditions — Acute Lung Injury | interventions — voxelotor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Voxelotor Arm (Experimental): 500 mg of Voxelotor two times a day (for a total daily dose of 1000 mg per day) for 5 days. This dose may increase to a total maximum daily dose of 1500 mg (500 mg three times a day), if subject tolerates the initial dose as determined by study doctor.
  Interventions: Drug: Voxelotor

INTERVENTIONS:
Drug: Voxelotor — 500 mg of voxelotor will be administered two times a day (for a total daily dose of 1000 mg per day) for 5 days. This dose may increase to a total maximum daily dose of 1500 mg (500 mg three times a day) if subject tolerates initial dose as determined by Principal Investigator (PI).
  Other Names: Oxbryta®

SUMMARY:
The purpose of the study is to evaluate the efficacy of voxelotor for increasing oxygen saturation in 20 patients with hypoxemia. Specifically, the SpO2/FiO2 ratio will be compared before and after voxelotor use at rest and during exercise (ambulatory patients only).

The primary study objective is to evaluate the efficacy of voxelotor for increasing oxygen saturation in patients with hypoxic hypoxemia as a result of end-stage lung disease or acute lung injury.

The secondary objective is to evaluate the efficacy of voxelotor on allowing de-escalation of supplemental oxygen support.

DETAILED DESCRIPTION:
Purpose of the study: Primary study objective is to evaluate the efficacy of voxelotor for increasing oxygen saturation in patients with hypoxic hypoxemia as a result of end-stage lung disease or acute lung injury.

Design and Procedures: The day after obtaining written informed consent, 20 patients will receive 500 mg of voxelotor two times a day (for a total daily dose of 1000 mg per day) for 5 days This dose may increase to a total maximum daily dose of 1500 mg (500 mg three times a day) if subject tolerates initial dose as determined by Principal Investigator (PI).

Physiological data at screening, baseline, study day 1 - 5, and up to two days post voxelotor administration will be recorded from standard of care with the only exception being SpO2/FiO2 (S/F) ratio measurements, which will be obtained at the same intervals but by the qualified and delegated study staff or medical team through the use of an FiO2 weaning maneuver.

Study subjects will be asked to rate their dyspnea symptoms daily to record their perceived shortness of breath.

Blood samples will be collected the day prior to voxelotor administration, on study days 1 - 5, and on the 2 wash-out days following voxelotor administration.

ELIGIBILITY:
Inclusion Criteria:

* Oxygen dependency due to an end-staged lung disease (pre-lung transplant population) or ALI/acute lung injury (for example but not limited to primary allograft dysfunction, infectious pneumonia, aspiration, non-cardiogenic pulmonary edema). ALI will be defined as per Berlin criteria with a P/F ratio <100 denoting severe ARDS, <200 denoting moderate and <300 mild ARDS. ALI and mild ARDS are considered synonymous. In the event of inability to obtain arterial blood gas analysis to calculate a P/F ratio, we will consider a range of patients requiring standard nasal cannulae flowing at 6l/min to maintain SaO2 >90% as ALI, and Salter High -Flow nasal cannulae at 12-15l/min in order to maintain SaO2>85% as severe ARDS.
* At least 48 hours of stable, increased oxygen requirement or ventilatory support prior to the start of drug administration if consented.

Exclusion Criteria:

* Minors (<18 years)
* Pre-existing congestive cardiac failure (NYHA III or IV)
* Medically significant, non-revascularized coronary artery disease
* Inability to obtain informed consent from LAR
* Pregnancy
* Incarcerated individual.
* Failure of another vital organ.
* Severe hepatic impairment (Childs-Pugh C) or liver enzymes > 4x upper limit of normal (ULN) at screening.
* Unstable acute kidney injury/rising creatinine.
* Chronic neuromuscular disease requiring mechanical ventilation
* Not anticipated to survive >48 hours
* Limited therapeutic goals (do not resuscitate, etc.)
* History of Pulmonary Embolism (PE)
* Requires treatment with Fluconazole or other moderate and strong CYP3A4 inhibitors listed in section 5.6
* A patient with active bleeding complications requiring more than 1 unit of blood transfusion per day, as the PK and PD of Voxelotor in the setting of blood loss and blood transfusion is unknown.
* Participated in another clinical trial of an investigational drug (or medical device) within 30 days or 5-half-lives, whichever is longer, prior to consent, or is currently participating in another trial of an investigational or marketed drug (or medical device)
* Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
* Any condition or concomitant medication that confounds the ability to interpret data from the study or safely use Voxelotor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Welsby, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Voxelotor Arm
Started | 3
Completed | 2
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Voxelotor Arm
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in SpO2/FiO2 (S/F) Ratio From Baseline to 2 Days After Initiation of Voxelotor Treatment
Description: SpO2 (oxygen saturation) is the percentage of oxygen in the blood. The fraction of inspired oxygen (FiO2) is the concentration of oxygen a person inhales.
Time Frame: baseline to 2 days after initiation of voxelotor treatment
Population: Participants with data collected at both timepoints.
Measure: Median (Standard Deviation); unit: SpO2/FiO2
Arm/Group | Voxelotor Arm
Number analyzed (Participants) | 2
SpO2/FiO2 | 0.105 (0.215)

2. Secondary Outcome: Change in SpO2/FiO2 (S/F) Ratio From Baseline to 5 Days After Initiation of Voxelotor Treatment
Description: as for outcome 1
Time Frame: baseline to 5 days after initiation of voxelotor treatment
Population: Participants with data collected at both timepoints.
Measure: Median (Standard Deviation); unit: SpO2/FiO2
Arm/Group | Voxelotor Arm
Number analyzed (Participants) | 2
SpO2/FiO2 | -0.01 (0.11)

ADVERSE EVENTS:
Time Frame: Participants will be followed for AEs from the time of voxelotor administration until 2 days after the last administration of voxelotor as defined by the wash out period.
Arm/Group | Voxelotor Arm
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voxelotor Arm (N=3)
Diarrhea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT05289570/Prot_SAP_000.pdf